CLINICAL TRIAL: NCT04658056
Title: The UK POST WATERStudy: UK Post-market Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue
Brief Title: UK Post-market Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP0002
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WATER AQUABEAM Robotic System cohort: WATER Study subjects previously-treated with Aquablation of the prostate with the AQUABEAM Robotic System for lower urinary tract symptoms associated with BPH.
- WATER TURPS cohort: WATER Study subjects previously-treated with standard transurethral resection of the prostate (TURP) for lower urinary tract symptoms associated with BPH.

SUMMARY:
A post-market, non-interventional, two-arm, long-term follow-up study of patients previously enrolled in the WATER Study (NCT02505919) - which was a prospective multi-centre randomized blinded study comparing Aquablation of the prostate with the AQUABEAM Robotic System with standard transurethral resection of the prostate (TURP) for the treatment of lower urinary tract symptoms (LUTS).

DETAILED DESCRIPTION:
The study is a post-market, non-interventional, two-arm, long-term follow-up study of patients previously enrolled in the WATER Study (NCT02505919) - which was a prospective multi-centre randomized blinded study comparing Aquablation of the prostate with the AQUABEAM Robotic System with standard transurethral resection of the prostate (TURP) for the treatment of lower urinary tract symptoms (LUTS). In POST WATER, up to 46 WATER Study subjects in the United Kingdom who were active on the study at 36 months will be invited to participate, across 3 clinical study sites in England and Wales. The study will consist of one follow-up time-point at 60 months (5 years) from the time of initial WATER Study treatment date.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was randomized and received treatment in the WATER Study.
2. Subject is mentally capable and willing to sign a study-specific informed consent form
3. Subject is willing and able to comply with all study requirements

Exclusion Criteria:

Dementia or psychiatric condition that prevents the participant from completing required follow up 2. Participating in another investigational study that could affect responses to the study assessments

Ages: 45 Years to 85 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The target patient population is subjects who were enrolled in the WATER Study (with symptomatic BPH) who were randomized to treatment with either the Aquablation procedure or TURP.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Long-term effectiveness as measured by IPSS at 60 months | 60 months following original surgical intervention
  International Prostate Symptom Score at 60 months as compared to baseline
Long-term safety as measured by adverse events at 60 months | 60 months following original surgical intervention
  The proportion of subjects with adverse events classified as Clavien-Dindo Grade 2 or higher or any grade 1 event resulting in persistent disability

OTHER OUTCOMES:
Reoperation or Re-intervention at 60 months | 60 months
  Reoperation or Re-intervention at 60 months
IPSS-QoL at 60 months | 60 months
  International Prostate Symptom Score Quality of Life sub-score
Qmax at 60 months | 60 months
  Uroflowmetry measurement of voided urine (in milliliters) per unit of time (in seconds)
PVR at 60 months | 60 months
  Post-void residual urine test
Erectile function at 60 months | 60 months
  IIEF-15 score
MSHQ-EjD at 60 months | 60 months
  Assessment of ejaculatory function/dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roehrborn, MD, Principal Investigator — UT Southwestern Medical; Peter Gilling, MD, Principal Investigator — Tauranga Urology Research Limited
Locations (1):
- Frimley Park Hospital, Camberley, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. Three-year outcomes after Aquablation therapy compared to TURP: results from a blinded randomized trial. Can J Urol. 2020 Feb;27(1):10072-10079. PMID 32065861
- [Result] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. Two-Year Outcomes After Aquablation Compared to TURP: Efficacy and Ejaculatory Improvements Sustained. Adv Ther. 2019 Jun;36(6):1326-1336. doi: 10.1007/s12325-019-00952-3. Epub 2019 Apr 26. PMID 31028614
- [Result] Pimentel MA, Yassaie O, Gilling P. Urodynamic Outcomes After Aquablation. Urology. 2019 Apr;126:165-170. doi: 10.1016/j.urology.2019.01.020. Epub 2019 Feb 2. PMID 30721737
- [Result] Gilling PJ, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Roehrborn C. Randomized Controlled Trial of Aquablation versus Transurethral Resection of the Prostate in Benign Prostatic Hyperplasia: One-year Outcomes. Urology. 2019 Mar;125:169-173. doi: 10.1016/j.urology.2018.12.002. Epub 2018 Dec 12. PMID 30552937
- [Result] Chughtai B, Thomas D. Pooled Aquablation Results for American Men with Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia in Large Prostates (60-150 cc). Adv Ther. 2018 Jun;35(6):832-838. doi: 10.1007/s12325-018-0722-0. Epub 2018 Jun 5. PMID 29873008